CLINICAL TRIAL: NCT02038036
Title: Randomized, Open Label, Multicenter Phase IIIb Study Evaluating the Efficacy and Safety of Ruxolitinib Versus Best Available Therapy in Patients With Polycythemia Vera Who Are Hydroxyurea Resistant or Intolerant (Response 2)
Brief Title: Ruxolitinib Efficacy and Safety in Patients With HU Resistant or Intolerant Polycythemia Vera vs Best Available Therapy.
Acronym: RESPONSE-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CINC424B2401
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Results first posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-06

CONDITIONS: Polycythemia Vera
Keywords: Polycythemia Vera; Hematologic Diseases; Myeloproliferative Disorders; Bone Marrow Diseases; Hydroxyurea; INC424; Ruxolitinib
MeSH Terms: conditions — Polycythemia Vera; Hematologic Diseases; Myeloproliferative Disorders; Bone Marrow Diseases | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ruxolitinib (Experimental): Ruxolitinib was administered at a starting dose of 10 mg twice a day (bid). Dose was adjusted based on efficacy and safety parameters up to a maximum dose of 25 mg bid.
  Interventions: Drug: Ruxolitinib
- Best Available Therapy (BAT) (Active Comparator): Best Available Therapy as selected by the investigator from: Hydroxyurea, Pegylated-Interferon (IFN/PEG-IFN), pipobroman, anagrelide, IMIDs, or observation. Participants randomized to BAT who did not respond by Week 28 were eligible to crossover and start treatment with ruxolitinib.
  Interventions: Drug: Best Available Therapy

INTERVENTIONS:
Drug: Best Available Therapy — Best Available Therapy as selected by the investigator from: Hydroxyurea, Pegylated-Interferon (IFN/PEG-IFN), pipobroman, anagrelide, IMIDs, or observation. Participants randomized to BAT who did not respond by Week 28 were eligible to crossover and start treatment with ruxolitinib.
  Other Names: BAT
  Arms: Best Available Therapy (BAT)
Drug: Ruxolitinib — Ruxolitinib was administered at a starting dose of 10 mg twice a day (bid). Dose was adjusted based on efficacy and safety parameters up to a maximum dose of 25 mg bid.
  Other Names: INC424
  Arms: Ruxolitinib

SUMMARY:
This study compared the efficacy and safety of ruxolitinib to Best Available Therapy (BAT) in patients with polycythemia vera (PV) who were hydroxyurea (HU) resistant or intolerant and did not have a palpable spleen.

DETAILED DESCRIPTION:
This was a prospective, multi-center, open-label, randomized, Phase IIIb study evaluating efficacy and safety of ruxolitinib versus BAT as selected by the Investigator in patients with PV who are resistant to, or intolerant of HU.

The study comprised of the following periods:

Screening Period (up to 5 weeks: Day -35 to Day -1): Screening evaluations were performed at one or more clinic visits, and reviewed to determine eligibility before the patient was randomized in the study.

Core Treatment Period (Day 1 to Week 80):

Patients were randomized in 1:1 ratio to either treatment group (ruxolitinib or BAT) and were to be treated with their randomized treatment.

Crossover Treatment Period (Week 28 or after) for BAT patients only:

Patients randomized to BAT who did not respond by Week 28 were eligible to crossover and start treatment with ruxolitinib. Patients crossing over on or after Week 28 had to complete all assessments for the End of Treatment (EoT) visit of the Core Treatment Period followed by the assessments in Cross-over visit evaluation schedule.

Extended Treatment Period (Week 80 to Week 260):

Patients receiving ruxolitinib at Week 80 (including patients who have crossed over from BAT) were eligible to continue up to Week 260 in the Extended Treatment Period. Patients continued the ruxolitinib dose that they received at Week 80. Patients who received BAT at Week 80 were not eligible to enter the Extended Treatment Period and had to have the EoT visit at Week 80 and an End of study (EoS) visit 30 days after the EoT visit.

Follow-up Period:

Patients were followed for safety during 30 days after the last dose of study drug and EoS visit assessments were performed post 30 days after the last dose of study drug. Patients who completed EoT (Week 80 for patients who received BAT, Week 260 for patients who received ruxolitinib or from the time of premature discontinuation) were to be followed-up for every 3 months for survival till the end of the study.

ELIGIBILITY:
Inclusion Criteria:

Confirmed diagnosis of PV according to the 2008 World Health Organization criteria, Non-palpable spleen, Phlebotomy dependent, Resistant to or intolerant of hydroxyurea, ECOG performance status of 0, 1 or 2.

Exclusion Criteria:

Inadequate liver or renal function, Significant bacterial, fungal, parasitic, or viral infection requiring treatment, Active malignancy within the past 5 years, excluding specific skin cancers, Previously received treatment with a JAK inhibitor, Being treated with any investigational agent, Women who are pregnant or nursing.

Other inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2014-03-25 (Actual); Primary Completion 2015-09-29 (Actual); Study Completion 2020-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (46):
- Novartis Investigative Site, Herston, Queensland, Australia
- Belgium (2):
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Leuven
- Novartis Investigative Site, Toronto, Ontario, Canada
- France (7):
  - Novartis Investigative Site, Bayonne, Bayonne Cedex
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
- Germany (9):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, Ulm
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Kaposvár
- India (2):
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Vellore, Tamil Nadu
- Israel (3):
  - Novartis Investigative Site, Nahariya
  - Novartis Investigative Site, Netanya
  - Novartis Investigative Site, Tel Aviv
- Italy (7):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Rome, Lazio
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Varese, VA
- Novartis Investigative Site, Seoul, South Korea
- Spain (8):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Las Palmas de Gran Canaria, Las Palmas de G.C
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Madrid
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Talas / Kayseri

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Passamonti F, Palandri F, Saydam G, Callum J, Devos T, Guglielmelli P, Vannucchi AM, Zor E, Zuurman M, Gilotti G, Zhang Y, Griesshammer M. Ruxolitinib versus best available therapy in inadequately controlled polycythaemia vera without splenomegaly (RESPONSE-2): 5-year follow up of a randomised, phase 3b study. Lancet Haematol. 2022 Jul;9(7):e480-e492. doi: 10.1016/S2352-3026(22)00102-8. Epub 2022 May 18. PMID 35597252
- [Derived] Kiladjian JJ, Guglielmelli P, Griesshammer M, Saydam G, Masszi T, Durrant S, Passamonti F, Jones M, Zhen H, Li J, Gadbaw B, Perez Ronco J, Khan M, Verstovsek S. Efficacy and safety of ruxolitinib after and versus interferon use in the RESPONSE studies. Ann Hematol. 2018 Apr;97(4):617-627. doi: 10.1007/s00277-017-3225-1. Epub 2018 Feb 2. PMID 29396713
- [Derived] Passamonti F, Griesshammer M, Palandri F, Egyed M, Benevolo G, Devos T, Callum J, Vannucchi AM, Sivgin S, Bensasson C, Khan M, Mounedji N, Saydam G. Ruxolitinib for the treatment of inadequately controlled polycythaemia vera without splenomegaly (RESPONSE-2): a randomised, open-label, phase 3b study. Lancet Oncol. 2017 Jan;18(1):88-99. doi: 10.1016/S1470-2045(16)30558-7. Epub 2016 Dec 2. PMID 27916398

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized in 48 centers across 12 countries: Australia (1), Belgium (2), Canada (1), France (7), Germany (9), Hungary (3), India (2), Israel (3), Italy (7), South Korea (2), Spain (9) and Turkey (2)
Pre-assignment Details: Participants were randomized in a 1:1 ratio either to Ruxolitinib or Best available Therapy (BAT). Randomization was stratified by patients who were resistant to or intolerant of Hydroxyurea (HU).
Groups:
- Ruxolitinib: Ruxolitinib at a starting dose of 10 mg twice a day (bid). Dose was adjusted based on efficacy and safety parameters up to a maximum dose of 25 mg bid
Period: Core Study
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Started | 74 | 75
Full Analysis Set (comprised of all patients to whom study treatment was assigned by randomization.) | 74 | 75
Crossover Set (consisted of all patients randomized to the BAT arm, who crossed over and received at least one dose of ruxolitinib.) | 0 | 58
Completed | 59 | 61
Not Completed | 15 | 14
Not completed — Adverse Event | 7 | 7
Not completed — Death | 1 | 1
Not completed — Disease progression | 2 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Subject/guardian decision | 0 | 1
Not completed — Withdrawal by Subject | 3 | 1
Period: Crossover Period
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Started | 0 | 58 (58 participants were eligible to crossover to the ruxolitinib arm)
Completed | 0 | 38
Not Completed | 0 | 20
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Adverse Event | 0 | 9
Not completed — Death | 0 | 2
Not completed — Disease progression | 0 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ruxolitinib | Best Available Therapy (BAT) | Total
Number analyzed (Participants) | 74 | 75 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (11.31) | 66.0 (11.12) | 64.4 (11.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 28 | 63
  Male | 39 | 47 | 86
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 67 | 66 | 133
  Asian | 4 | 5 | 9
  Other | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Hematocrit (Hct) Control at Week 28
Description: Proportion of patients achieving Hct control at Week 28 was defined by the absence of phlebotomy eligibility starting at Week 8 and continuing through Week 28, with no more than one phlebotomy eligibility occurring post randomization and prior to Week 8.
  Phlebotomy eligibility was defined by:
  * Confirmed Hct > 45% that is at least 3 percentage points higher than the Hct obtained at Baseline Or
  * Confirmed Hct > 48% The confirmation occurred 2 to 14 days subsequent to the initial observation.
Time Frame: Week 28
Population: Full Analysis Set (FAS) included all participants to whom study treatment was assigned by randomization and had valid measurements for the outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 74 | 75
Participants | 46 | 14

2. Secondary Outcome: Number of Participants Achieving a Complete Hematological Remission at Week 28
Description: Proportion of patients achieving a complete hematological remission at Week 28 was defined by:
  * Hct control at Week 28 defined by the absence of phlebotomy eligibility starting at Week 8 and continuing through Week 28, with no more than one phlebotomy eligibility occurring post randomization and prior to Week 8, and
  * WBC < 10 x109/L at Week 28, and
  * Platelets ≤ 400 x 109/L at Week 28
Time Frame: Week 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 74 | 75
Participants | 17 | 4

3. Secondary Outcome: Number of Participants Achieving a Hematocrit (Hct) Control at Week 52 and Week 80
Description: Proportion of patients achieving a Hct control at Week 52 was defined by the absence of phlebotomy eligibility starting at Week 8 and continuing through Week 52, and no more than one phlebotomy eligibility occurring post randomization and prior to Week 8
  - Endpoint for Week 80 was defined, similarly.
Time Frame: Week 52 and 80
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 74 | 75
Participants
  Week 52 | 44 | 5
  Week 80 | 35 | 2

4. Secondary Outcome: Number of Participants Achieving a Complete Hematological Remission at Week 52 and Week 80
Description: Proportion of patients achieving a complete hematological remission at Week 52, was defined by:
  * Hct control at Week 52, as defined by the absence of phlebotomy eligibility starting at Week 8 and continuing through Week 52 with no more than one phlebotomy eligibility occurring post randomization and prior to Week 8, and
  * White Blood Count (WBC) < 10 x10^9/L at Week 52, and
  * Platelets ≤ 400 x 10^9/L at Week 52
  * Endpoint for Week 80 was defined, similarly.
Time Frame: Week 52 and 80
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 74 | 75
Participants
  Week 52 | 17 | 3
  Week 80 | 18 | 2

5. Secondary Outcome: Number of Participants With Phlebotomies Over Time
Description: Phlebotomy eligibility was defined by Confirmed Hct > 45% that is at least 3 percentage points higher than the Hct obtained at Baseline Or Confirmed Hct > 48%. The confirmation occurred 2 to 14 days subsequent to the initial observation.
Time Frame: Baseline to Week 260
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 74 | 75
Participants
  Phlebotomy frequency: >0 - <=2 | 12 | 29
  Phlebotomy frequency: >2 - <=4 | 7 | 17
  Phlebotomy frequency: >4 - <=6 | 4 | 2
  Phlebotomy frequency: >6 - <=8 | 0 | 1

6. Secondary Outcome: Change From Baseline in Hematocrit (Hct) at Each Visit
Description: Hematocrit is the volume percentage of red blood cells (RBC) in the blood.
Time Frame: Baseline, Week 4, 8, 12, 16, 20, 24, 28, 40, 52, 66, 80, 92, 104, 117, 130, 143, 156, 169, 182, 195, 208, 221, 234, 247 and 260
Population: Full Analysis Set (FAS) included all participants to whom study treatment was assigned by randomization and had valid measurements for the outcome measure. Data after crossover for participants randomized to BAT are reported as separate outcome measure.
Measure: Mean (Standard Deviation); unit: volume percentage of RBC in blood
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 74 | 75
volume percentage of RBC in blood
  Week 4: number analyzed (Participants) | 67 | 69
  Week 4 | -0.65 (2.943) | 1.25 (2.994)
  Week 8: number analyzed (Participants) | 67 | 71
  Week 8 | -1.22 (3.634) | 1.63 (3.344)
  Week 12: number analyzed (Participants) | 65 | 71
  Week 12 | -2.33 (4.581) | 1.70 (3.485)
  Week 16: number analyzed (Participants) | 66 | 70
  Week 16 | -3.25 (4.179) | 1.83 (3.439)
  Week 20: number analyzed (Participants) | 68 | 68
  Week 20 | -3.05 (4.307) | 1.45 (3.984)
  Week 24: number analyzed (Participants) | 64 | 63
  Week 24 | -2.85 (4.094) | 1.52 (2.934)
  Week 28: number analyzed (Participants) | 65 | 67
  Week 28 | -2.60 (4.101) | 2.09 (3.852)
  Week 40: number analyzed (Participants) | 67 | 24
  Week 40 | -2.77 (4.538) | 2.05 (4.587)
  Week 52: number analyzed (Participants) | 65 | 16
  Week 52 | -2.49 (4.445) | 1.68 (4.854)
  Week 66: number analyzed (Participants) | 63 | 11
  Week 66 | -3.06 (4.573) | 2.73 (2.922)
  Week 80: number analyzed (Participants) | 61 | 6
  Week 80 | -3.20 (3.886) | 0.62 (4.436)
  Week 92: number analyzed (Participants) | 64 | 0
  Week 92 | -2.91 (4.203) |
  Week 104: number analyzed (Participants) | 61 | 0
  Week 104 | -3.19 (4.314) |
  Week 117: number analyzed (Participants) | 63 | 0
  Week 117 | -2.86 (4.540) |
  Week 130: number analyzed (Participants) | 63 | 0
  Week 130 | -3.13 (4.263) |
  Week 143: number analyzed (Participants) | 60 | 0
  Week 143 | -3.50 (3.463) |
  Week 156: number analyzed (Participants) | 61 | 0
  Week 156 | -3.54 (4.005) |
  Week 169: number analyzed (Participants) | 58 | 0
  Week 169 | -3.57 (4.477) |
  Week 182: number analyzed (Participants) | 58 | 0
  Week 182 | -2.94 (4.428) |
  Week 195: number analyzed (Participants) | 58 | 0
  Week 195 | -3.36 (4.515) |
  Week 208: number analyzed (Participants) | 55 | 0
  Week 208 | -3.23 (4.150) |
  Week 221: number analyzed (Participants) | 54 | 0
  Week 221 | -3.55 (4.413) |
  Week 234: number analyzed (Participants) | 56 | 0
  Week 234 | -3.31 (4.621) |
  Week 247: number analyzed (Participants) | 52 | 0
  Week 247 | -3.45 (4.053) |
  Week 260: number analyzed (Participants) | 40 | 0
  Week 260 | -2.93 (3.799) |

7. Secondary Outcome: Change From Baseline in Hematocrit (Hct) at Each Scheduled Visit After Crossover in Participants Randomized to BAT Who Cross Over to Ruxolitinib
Description: Hematocrit is the percentage of red blood cells (RBC) in the blood.
Time Frame: Baseline (last assessment before cross over), Week 4, 8, 12, 16, 20, 24, 28, 40, 52, 64, 76, 89, 102, 115, 128, 141, 154, 167, 180, 193, 206, 219 and 232 after cross-over
Population: Cross-over set consisted of all participants randomized to the BAT arm, who crossed over and received at least one dose of ruxolitinib.
Measure: Mean (Standard Deviation); unit: Volume percentage of RBC in blood
Groups:
- All Crossover Patients: Participants randomized to the BAT arm, who crossed over and received at least one dose of ruxolitinib
Arm/Group | All Crossover Patients
Number analyzed (Participants) | 58
Volume percentage of RBC in blood
  Week +4: number analyzed (Participants) | 57
  Week +4 | -2.44 (3.394)
  Week +8: number analyzed (Participants) | 52
  Week +8 | -4.24 (5.322)
  Week +12: number analyzed (Participants) | 54
  Week +12 | -5.73 (6.597)
  Week +16: number analyzed (Participants) | 53
  Week +16 | -6.27 (7.101)
  Week +20: number analyzed (Participants) | 54
  Week +20 | -5.76 (6.563)
  Week +24: number analyzed (Participants) | 52
  Week +24 | -5.29 (6.518)
  Week +28: number analyzed (Participants) | 51
  Week +28 | -6.04 (5.825)
  Week +40: number analyzed (Participants) | 53
  Week +40 | -6.06 (6.301)
  Week +52: number analyzed (Participants) | 49
  Week +52 | -5.91 (6.399)
  Week +64: number analyzed (Participants) | 50
  Week +64 | -7.06 (6.051)
  Week +76: number analyzed (Participants) | 48
  Week +76 | -6.16 (6.247)
  Week +89: number analyzed (Participants) | 48
  Week +89 | -6.79 (6.046)
  Week +102: number analyzed (Participants) | 47
  Week +102 | -6.21 (6.599)
  Week +115: number analyzed (Participants) | 48
  Week +115 | -7.04 (6.103)
  Week +128: number analyzed (Participants) | 46
  Week +128 | -7.41 (6.812)
  Week +141: number analyzed (Participants) | 41
  Week +141 | -7.00 (6.310)
  Week +154: number analyzed (Participants) | 30
  Week +154 | -7.06 (7.000)
  Week +167: number analyzed (Participants) | 29
  Week +167 | -7.44 (7.426)
  Week +180: number analyzed (Participants) | 37
  Week +180 | -7.51 (7.298)
  Week +193: number analyzed (Participants) | 38
  Week +193 | -7.16 (5.331)
  Week +206: number analyzed (Participants) | 39
  Week +206 | -7.09 (5.742)
  Week +219: number analyzed (Participants) | 35
  Week +219 | -6.95 (5.936)
  Week +232: number analyzed (Participants) | 33
  Week +232 | -7.51 (5.880)

8. Secondary Outcome: Spleen Length by Visit
Description: Spleen length was assessed by manual palpation at every study visit.
Time Frame: Week 4, 8, 12, 16, 20, 24, 28, 40, 52, 66, 80, 92, 104, 117, 130, 143, 156, 169, 182, 195, 208, 221, 234, 247 and 260
Population: Full Analysis Set (FAS) included all participants to whom study treatment was assigned by randomization and had valid measurements for the outcome measure. Data after crossover for participants randomized to BAT were not collected.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 74 | 75
cm
  Week 4: number analyzed (Participants) | 71 | 73
  Week 4 | 0.00 (0.000) | 0.04 (0.351)
  Week 8: number analyzed (Participants) | 71 | 71
  Week 8 | 0.00 (0.000) | 0.01 (0.119)
  Week 12: number analyzed (Participants) | 69 | 70
  Week 12 | 0.00 (0.000) | 0.01 (0.120)
  Week 16: number analyzed (Participants) | 69 | 70
  Week 16 | 0.00 (0.000) | 0.23 (1.010)
  Week 20: number analyzed (Participants) | 70 | 67
  Week 20 | 0.00 (0.000) | 0.13 (0.716)
  Week 24: number analyzed (Participants) | 68 | 64
  Week 24 | 0.00 (0.000) | 0.09 (0.555)
  Week 28: number analyzed (Participants) | 70 | 67
  Week 28 | 0.00 (0.000) | 0.20 (0.909)
  Week 40: number analyzed (Participants) | 70 | 23
  Week 40 | 0.01 (0.120) | 0.52 (1.473)
  Week 52: number analyzed (Participants) | 69 | 15
  Week 52 | 0.06 (0.482) | 0.07 (0.258)
  Week 66: number analyzed (Participants) | 68 | 10
  Week 66 | 0.00 (0.000) | 0.00 (0.000)
  Week 80: number analyzed (Participants) | 66 | 5
  Week 80 | 0.03 (0.246) | 0.00 (0.000)
  Week 92: number analyzed (Participants) | 67 | 0
  Week 92 | 0.00 (0.000) |
  Week 104: number analyzed (Participants) | 63 | 0
  Week 104 | 0.05 (0.378) |
  Week 117: number analyzed (Participants) | 66 | 0
  Week 117 | 0.12 (0.985) |
  Week 130: number analyzed (Participants) | 66 | 0
  Week 130 | 0.18 (1.162) |
  Week 143: number analyzed (Participants) | 61 | 0
  Week 143 | 0.08 (0.458) |
  Week 156: number analyzed (Participants) | 65 | 0
  Week 156 | 0.05 (0.372) |
  Week 169: number analyzed (Participants) | 63 | 0
  Week 169 | 0.05 (0.378) |
  Week 182: number analyzed (Participants) | 62 | 0
  Week 182 | 0.05 (0.381) |
  Week 195: number analyzed (Participants) | 60 | 0
  Week 195 | 0.00 (0.000) |
  Week 208: number analyzed (Participants) | 58 | 0
  Week 208 | 0.00 (0.000) |
  Week 221: number analyzed (Participants) | 60 | 0
  Week 221 | 0.02 (0.129) |
  Week 234: number analyzed (Participants) | 59 | 0
  Week 234 | 0.00 (0.000) |
  Week 247: number analyzed (Participants) | 54 | 0
  Week 247 | 0.02 (0.136) |
  Week 260: number analyzed (Participants) | 42 | 0
  Week 260 | 0.10 (0.617) |

9. Secondary Outcome: Change From Baseline in Eastern Cooperative Oncology Group (ECOG) Performance Status to Week 28
Description: The ECOG scale of performance status described the level of functioning of participants in terms of their ability to care for themselves, daily activity, and physical ability. The ECOG performance was recorded as per ECOG performance status grades ranging from 0 (fully active, able to carry on all pre-disease performance without restriction) to 5 (dead).
Time Frame: Baseline and Week 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 74 | 75
Participants
  Grade 0 at baseline: number analyzed (Participants) | 53 | 56
  Grade 0 at baseline: 0: Fully active, able to carry on all pre-disease performance without restriction | 49 | 17
  Grade 0 at baseline: 1: Restricted in physically strenuous activity and able to carry out light or sedentary work | 2 | 1
  Grade 0 at baseline: 2: Ambulatory and capable of all self-care but unable to carry out any work activities | 0 | 0
  Grade 0 at baseline: 3: Capable of only limited self-care, confined to bed or chair more than 50% of waking hours | 0 | 0
  Grade 0 at baseline: 4: Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair | 0 | 0
  Grade 0 at baseline: Missing | 2 | 38
  Grade 1 at baseline: number analyzed (Participants) | 21 | 19
  Grade 1 at baseline: 0: Fully active, able to carry on all pre-disease performance without restriction | 9 | 1
  Grade 1 at baseline: 1: Restricted in physically strenuous activity and able to carry out light or sedentary work | 10 | 5
  Grade 1 at baseline: 2: Ambulatory and capable of all self-care but unable to carry out any work activities | 1 | 0
  Grade 1 at baseline: 3: Capable of only limited self-care, confined to bed or chair more than 50% of waking hours | 0 | 0
  Grade 1 at baseline: 4: Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair | 0 | 0
  Grade 1 at baseline: Missing | 1 | 13

10. Secondary Outcome: Number of Participants Achieving a Partial Remission Based on the European Leukemia Net (ELN) and International Working Group for Myelofibrosis Research and Treatment (IWG-MRT) Criteria at Week 28
Description: Proportion of patients achieving a partial remission at Week 28, based on the ELN and IWG-MRT criteria, as defined by:
  * Myeloproliferative Neoplasm Symptom Assessment Form Total Symptom Score (MPN-SAF TSS) score reduction of greater than or equal to 10 points from baseline to Week 28, and
  * Hct control defined by the absence of phlebotomy eligibility starting at Week 8 and continuing through Week 28, with no more than one phlebotomy eligibility occurring post randomization and prior to Week 8, and
  * WBC < 10 x10^9/L at Week 28, and
  * Platelets ≤ 400 x 10^9/L at Week 28, and
  * No palpable spleen at Week 28, and
  * No hemorrhagic or thrombotic events, and
  * No transformation into post-PV myelofibrosis, myelodysplastic syndrome (IWG-MRT criteria) or acute leukemia (WHO criteria).
Time Frame: Week 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 74 | 75
Participants | 7 | 0

11. Secondary Outcome: Number of Participants Who Achieved Partial Remission Based on the European Leukemia Net (ELN) and International Working Group for Myelofibrosis Research and Treatment (IWG-MRT) Criteria at Week 52 and Week 80
Description: Proportion of patients who achieved partial remission at Week 52 based on the ELN and IWG-MRT criteria, as defined by:
  * MPN-SAF TSS score reduction of greater than or equal to 10 points from baseline to Week 52 and
  * Hct control defined by the absence of phlebotomy eligibility starting at Week 8 and continuing through Week 52 with no more than one phlebotomy eligibility occurring post randomization and prior to Week 8, and
  * WBC < 10 x109/L at Week 52 and
  * Platelets ≤ 400 x 109/L at Week 52 and
  * No palpable spleen at Week 52 and
  * No hemorrhagic or thrombotic events, and
  * No transformation into post-PV myelofibrosis, myelodysplastic syndrome (IWG-MRT criteria) or acute leukemia (WHO criteria).
  * Endpoint for Week 80 was defined, similarly.
Time Frame: Week 52 and 80
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 74 | 75
Participants
  Week 52 | 5 | 0
  Week 80 | 4 | 0

12. Secondary Outcome: Number of Participants Achieving a Hematocrit (Hct) Control at Week 104, Week 156, Week 208 and Week 260.
Description: Proportion of patients achieving a Hct control at Week 104 as defined by the absence of phlebotomy eligibility starting at Week 8 and continuing through Week 104 and with no more than one phlebotomy eligibility occurring post randomization and prior to Week 8 Endpoint for Week 156, Week 208 and Week 260 were defined, similarly.
Time Frame: From Week 8 to Week 104, 156, 208 and 260
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 74
Participants
  Week 104: number analyzed (Participants) | 34
  Week 104: HU Resistant | 9
  Week 104: HU Intolerant | 25
  Week 156: number analyzed (Participants) | 30
  Week 156: HU Resistant | 9
  Week 156: HU Intolerant | 21
  Week 208: number analyzed (Participants) | 25
  Week 208: HU Resistant | 7
  Week 208: HU Intolerant | 18
  Week 260: number analyzed (Participants) | 16
  Week 260: HU Resistant | 4
  Week 260: HU Intolerant | 12

13. Secondary Outcome: Number of Participants Achieving a Complete Hematological Remission at Week 104, Week 156, Week 208 and Week 260
Description: Proportion of patients achieving a complete hematological remission at Week 104 as defined by Hct control defined by the absence of phlebotomy eligibility starting at Week 8 and continuing through Week 104, with no more than one phlebotomy eligibility occurring post randomization and prior to Week 8, and
  * WBC < 10 x10^9/L at Week 104, and
  * Platelets ≤ 400 x 10^9/L at Week 104 Endpoint for Week 156, Week 208 and Week 260 were defined, similarly.
Time Frame: From Week 8 to Week 104, 156, 208 and 260
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 74
Participants
  Week 104 | 15
  Week 156 | 19
  Week 208 | 11
  Week 260 | 9

14. Secondary Outcome: Number of Participants Who Achieved Partial Remission Based on the European Leukemia Net (ELN) and International Working Group for Myelofibrosis Research and Treatment (IWG-MRT) Criteria at Week 104, Week 156, Week 208 and Week 260.
Description: Proportion of patients who achieved partial remission at Week 104, based on the ELN and IWG-MRT criteria, as defined by:
  * MPN-SAF TSS score reduction of greater than or equal to 10 points from baseline to Week 104, and
  * Hct control defined by the absence of phlebotomy eligibility starting at Week 8 and continuing through Week 104, with no more than one phlebotomy eligibility occurring post-randomization and prior to Week 8, and
  * WBC < 10 x10^9/L at Week 104, and
  * Platelets ≤ 400 x 10^9/L at Week 104, and
  * No palpable spleen at Week 104, and
  * No hemorrhagic or thrombotic events, and
  * No transformation into post-PV myelofibrosis, myelodysplastic syndrome (IWG-MRT criteria) or acute leukemia (WHO criteria) Endpoint for Week 156, Week 208 and Week 260 are defined, similarly.
Time Frame: From Week 8 to Week 104, 156, 208 and 260
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 74
Participants
  Week 104 | 4
  Week 156 | 9
  Week 208 | 4
  Week 260 | 0

15. Secondary Outcome: Number of Participants With Transformation Free Survival Events
Description: Transformation-free survival is defined as one of the following:
  1. Myelofibrosis (MF) as evidenced by bone marrow biopsy, or
  2. Acute leukemia as evidenced by bone marrow blast counts of at least 20%, or peripheral blast counts of at least 20% lasting at least 2 weeks.
  3. Death due to any cause during treatment period
Time Frame: Week 260 (ruxolitinib arm) and Week 80 (BAT arm)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 74 | 75
Participants | 4 | 3

16. Secondary Outcome: Number of Participants With Overall Survival (OS) Events
Description: Overall survival (OS) event is defined as death due to any cause. OS events were counted in the BAT arm, irrespective of whether participants crossed over to receive ruxolitinib when the event occurred.
Time Frame: up to Week 260
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 74 | 75
Participants | 3 | 6

17. Secondary Outcome: Change From Baseline in Myeloproliferative Neoplasm Symptom Assessment Form Total Symptom Score (MPN-SAF TSS)
Description: The MPN-SAF TSS is a disease specific questionnaire comprised of 10 items that measures fatigue related to MPN disease and the severity of nine of the most prevalent associated symptoms. Each item is scored on a scale ranging from 0 (no fatigue/absent) to 10 (As bad as you can imagine/worst imaginable).The MPN-SAF TSS is computed as the average of the observed items multiplied by 10 to achieve a 0-to-100 scale. The MPN-SAF TSS thus has a possible score range of 0 to 100 where a decrease indicates improvement.
Time Frame: Baseline, Week 4, 8, 16, 28, 40, 52, 80, 92, 104, 117, 130, 143, 156, 169, 182, 195, 208, 221, 234 and 247
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 74 | 75
Score on a scale
  Week 4: number analyzed (Participants) | 68 | 70
  Week 4 | -8.43 (12.341) | 0.40 (12.586)
  Week 8: number analyzed (Participants) | 68 | 69
  Week 8 | -9.86 (12.210) | 1.37 (12.046)
  Week 16: number analyzed (Participants) | 67 | 67
  Week 16 | -9.14 (13.980) | 1.41 (10.760)
  Week 28: number analyzed (Participants) | 65 | 23
  Week 28 | -10.29 (14.204) | 2.34 (13.047)
  Week 40: number analyzed (Participants) | 67 | 18
  Week 40 | -9.35 (14.027) | 0.10 (9.586)
  Week 52: number analyzed (Participants) | 70 | 13
  Week 52 | -8.63 (13.403) | 0.63 (9.334)
  Week 80: number analyzed (Participants) | 67 | 0
  Week 80 | -9.04 (13.520) |
  Week 92: number analyzed (Participants) | 64 | 0
  Week 92 | -7.69 (11.971) |
  Week 104: number analyzed (Participants) | 68 | 0
  Week 104 | -6.82 (13.297) |
  Week 117: number analyzed (Participants) | 64 | 0
  Week 117 | -6.76 (13.702) |
  Week 130: number analyzed (Participants) | 64 | 0
  Week 130 | -8.26 (16.234) |
  Week 143: number analyzed (Participants) | 64 | 0
  Week 143 | -8.56 (15.653) |
  Week 156: number analyzed (Participants) | 65 | 0
  Week 156 | -8.48 (15.081) |
  Week 169: number analyzed (Participants) | 64 | 0
  Week 169 | -7.65 (14.392) |
  Week 182: number analyzed (Participants) | 63 | 0
  Week 182 | -9.34 (14.675) |
  Week 195: number analyzed (Participants) | 61 | 0
  Week 195 | -7.57 (14.922) |
  Week 208: number analyzed (Participants) | 55 | 0
  Week 208 | -9.26 (16.347) |
  Week 221: number analyzed (Participants) | 55 | 0
  Week 221 | -7.20 (16.054) |
  Week 234: number analyzed (Participants) | 57 | 0
  Week 234 | -7.50 (15.922) |
  Week 247: number analyzed (Participants) | 51 | 0
  Week 247 | -7.82 (16.905) |

18. Secondary Outcome: Change From Baseline in Total Scores of MPN-SAF by Visit in Patients From BAT Group Who Cross Over to Ruxolitinib After Crossover
Description: as for outcome 17
Time Frame: Baseline (last assessment before cross over), Week 4, 8, 16, 24, 28, 40, 52, 92, 104, 117, 130, 143, 156, 169, 182, 195, 208, 221, 234 and 247 after cross-over
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Best Available Therapy (BAT): Participants randomized to the BAT arm, who crossed over and received at least one dose of ruxolitinib
Arm/Group | Best Available Therapy (BAT)
Number analyzed (Participants) | 58
Score on a scale
  Week +4: number analyzed (Participants) | 52
  Week +4 | -8.00 (10.532)
  Week +8: number analyzed (Participants) | 53
  Week +8 | -9.76 (11.543)
  Week +16: number analyzed (Participants) | 52
  Week +16 | -9.40 (12.040)
  Week +24: number analyzed (Participants) | 51
  Week +24 | -9.15 (12.738)
  Week +28: number analyzed (Participants) | 50
  Week +28 | -8.46 (12.212)
  Week +40: number analyzed (Participants) | 46
  Week +40 | -8.58 (13.302)
  Week +52: number analyzed (Participants) | 42
  Week +52 | -7.15 (14.392)
  Week 92: number analyzed (Participants) | 45
  Week 92 | -10.49 (13.902)
  Week 104: number analyzed (Participants) | 51
  Week 104 | -8.08 (16.288)
  Week 117: number analyzed (Participants) | 49
  Week 117 | -9.01 (14.708)
  Week 130: number analyzed (Participants) | 46
  Week 130 | -10.18 (15.740)
  Week 143: number analyzed (Participants) | 47
  Week 143 | -8.36 (17.030)
  Week 156: number analyzed (Participants) | 45
  Week 156 | -9.54 (14.573)
  Week 169: number analyzed (Participants) | 42
  Week 169 | -11.15 (14.305)
  Week 182: number analyzed (Participants) | 43
  Week 182 | -10.13 (16.113)
  Week 195: number analyzed (Participants) | 41
  Week 195 | -10.88 (14.357)
  Week 208: number analyzed (Participants) | 40
  Week 208 | -9.43 (15.360)
  Week 221: number analyzed (Participants) | 38
  Week 221 | -10.02 (15.986)
  Week 234: number analyzed (Participants) | 36
  Week 234 | -8.01 (14.404)
  Week 247: number analyzed (Participants) | 37
  Week 247 | -9.84 (14.979)

19. Secondary Outcome: Change From Baseline in Score as Per European Quality of Life 5-Dimension 5-level (EQ-5D-5L) Questionnaire
Description: EQ-5D-5L is a standardized instrument for measuring health outcomes in a wide range of health conditions and treatments. It consists of visual analogue scale (EQ VAS) which records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labeled 'Best imaginable health state' and 'worst imaginable health state'. The EQ VAS scores were anchored on 100 = the best health you can imagine and 0 = worst health you can imagine.
Time Frame: Baseline, Week 4, 8, 16, 28, 52, 80, 92, 104, 117, 130, 143, 156, 169, 182, 195, 208, 221, 234 and 247
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 74 | 75
Score on a scale
  Week 4: number analyzed (Participants) | 67 | 69
  Week 4 | 4.24 (11.661) | 0.04 (18.323)
  Week 8: number analyzed (Participants) | 66 | 67
  Week 8 | 7.62 (14.846) | -2.73 (16.097)
  Week 16: number analyzed (Participants) | 63 | 65
  Week 16 | 6.35 (17.946) | -3.12 (14.435)
  Week 28: number analyzed (Participants) | 63 | 25
  Week 28 | 7.56 (14.309) | 0.16 (15.201)
  Week 52: number analyzed (Participants) | 66 | 14
  Week 52 | 7.36 (13.996) | 2.50 (10.697)
  Week 80: number analyzed (Participants) | 64 | 0
  Week 80 | 4.50 (18.273) |
  Week 92: number analyzed (Participants) | 62 | 0
  Week 92 | 6.77 (18.948) |
  Week 104: number analyzed (Participants) | 64 | 0
  Week 104 | 6.25 (18.143) |
  Week 117: number analyzed (Participants) | 62 | 0
  Week 117 | 6.42 (15.130) |
  Week 130: number analyzed (Participants) | 61 | 0
  Week 130 | 7.70 (16.488) |
  Week 143: number analyzed (Participants) | 59 | 0
  Week 143 | 5.68 (17.332) |
  Week 156: number analyzed (Participants) | 62 | 0
  Week 156 | 4.74 (19.032) |
  Week 169: number analyzed (Participants) | 61 | 0
  Week 169 | 6.08 (18.717) |
  Week 182: number analyzed (Participants) | 60 | 0
  Week 182 | 7.68 (17.992) |
  Week 195: number analyzed (Participants) | 59 | 0
  Week 195 | 6.41 (18.239) |
  Week 208: number analyzed (Participants) | 53 | 0
  Week 208 | 7.94 (18.614) |
  Week 221: number analyzed (Participants) | 53 | 0
  Week 221 | 3.64 (19.866) |
  Week 234: number analyzed (Participants) | 54 | 0
  Week 234 | 5.48 (18.625) |
  Week 247: number analyzed (Participants) | 50 | 0
  Week 247 | 6.28 (17.854) |

20. Secondary Outcome: Change From Baseline in EQ-5D-5L VAS, by Visit in Patients From BAT Group Who Cross Over to Ruxolitinib After Crossover
Description: as for outcome 19
Time Frame: Baseline (last assessment before cross over), Week 4, 8, 16, 24, 28, 52, 92, 104, 117, 130, 143, 156, 169, 182, 195, 208, 221, 234 and 247 after cross-over
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Best Available Therapy (BAT)
Number analyzed (Participants) | 58
Score on a scale
  Week +4: number analyzed (Participants) | 52
  Week +4 | 4.54 (14.756)
  Week +8: number analyzed (Participants) | 52
  Week +8 | 4.62 (15.807)
  Week +16: number analyzed (Participants) | 52
  Week +16 | 6.58 (14.667)
  Week +24: number analyzed (Participants) | 50
  Week +24 | 6.38 (17.564)
  Week +28: number analyzed (Participants) | 50
  Week +28 | 5.26 (15.923)
  Week +52: number analyzed (Participants) | 41
  Week +52 | 4.71 (21.006)
  Week 92: number analyzed (Participants) | 45
  Week 92 | 8.09 (16.119)
  Week 104: number analyzed (Participants) | 50
  Week 104 | 6.48 (18.085)
  Week 117: number analyzed (Participants) | 49
  Week 117 | 4.92 (16.983)
  Week 130: number analyzed (Participants) | 46
  Week 130 | 4.87 (20.047)
  Week 143: number analyzed (Participants) | 47
  Week 143 | 3.19 (17.798)
  Week 156: number analyzed (Participants) | 46
  Week 156 | 2.65 (20.221)
  Week 169: number analyzed (Participants) | 41
  Week 169 | 4.59 (13.731)
  Week 182: number analyzed (Participants) | 42
  Week 182 | 2.71 (19.673)
  Week 195: number analyzed (Participants) | 40
  Week 195 | 5.65 (18.286)
  Week 208: number analyzed (Participants) | 40
  Week 208 | 5.35 (18.099)
  Week 221: number analyzed (Participants) | 38
  Week 221 | 7.71 (16.701)
  Week 234: number analyzed (Participants) | 37
  Week 234 | 5.30 (18.342)
  Week 247: number analyzed (Participants) | 36
  Week 247 | 4.14 (16.427)

21. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI) Questionnaire
Description: The Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI:SHP) is a six item questionnaire which intended to measure work and activity impairment associated with polycythemia vera. WPAI consisted of 6 questions (Q1=Employment status; Q2=Hours absent from work due to the polycythemia vera; Q3=Hours absent from work due to other reasons; Q4=Hours actually worked; Q5=Impact of the polycythemia vera on productivity while working; Q6=Impact of the polycythemia vera on productivity while doing regular daily activities other than work). Higher WPAI scores indicated greater activity impairment. Scores were multiplied by 100 to express in percentages.
  Percent work time missed due to problem (past 7 days) =Q2/(Q2+Q4) Percent impairment while working due to problem (past 7 days): Q5/10 Percent overall work impairment due to problem (past 7 says): Q2/(Q2+Q4)+[(1 Q2/(Q2+Q4))x(Q5/10)] Percent activity impairment due to problem (past 7 says): Q6/10
Time Frame: Baseline, Week 4, 8, 16, 28, 52 and 80
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 74 | 75
Percent
  Percent work time missed due to problem (past 7 days) Week 4: number analyzed (Participants) | 18 | 18
  Percent work time missed due to problem (past 7 days) Week 4 | -5.50 (18.425) | -0.40 (13.928)
  Percent work time missed due to problem (past 7 days) Week 8: number analyzed (Participants) | 15 | 16
  Percent work time missed due to problem (past 7 days) Week 8 | -4.88 (13.381) | -4.35 (20.820)
  Percent work time missed due to problem (past 7 days) Week 16: number analyzed (Participants) | 17 | 17
  Percent work time missed due to problem (past 7 days) Week 16 | 4.50 (35.948) | 4.79 (25.917)
  Percent work time missed due to problem (past 7 days) Week 28: number analyzed (Participants) | 17 | 4
  Percent work time missed due to problem (past 7 days) Week 28 | -5.85 (17.119) | -2.19 (9.852)
  Percent work time missed due to problem (past 7 days) Week 52: number analyzed (Participants) | 17 | 2
  Percent work time missed due to problem (past 7 days) Week 52 | -2.82 (30.770) | -8.33 (11.785)
  Percent work time missed due to problem (past 7 days) Week 80: number analyzed (Participants) | 15 | 0
  Percent work time missed due to problem (past 7 days) Week 80 | 1.87 (34.151) |
  Percent impairment while working due to problem (past 7 days) Week 4: number analyzed (Participants) | 21 | 18
  Percent impairment while working due to problem (past 7 days) Week 4 | -6.67 (23.310) | 0.00 (14.951)
  Percent impairment while working due to problem (past 7 days) Week 8: number analyzed (Participants) | 19 | 17
  Percent impairment while working due to problem (past 7 days) Week 8 | -13.16 (19.164) | -0.59 (13.449)
  Percent impairment while working due to problem (past 7 days) Week 16: number analyzed (Participants) | 20 | 17
  Percent impairment while working due to problem (past 7 days) Week 16 | -14.00 (21.374) | 4.12 (16.977)
  Percent impairment while working due to problem (past 7 days) Week 28: number analyzed (Participants) | 21 | 4
  Percent impairment while working due to problem (past 7 days) Week 28 | -14.29 (23.994) | -10.00 (14.142)
  Percent impairment while working due to problem (past 7 days) Week 52: number analyzed (Participants) | 20 | 2
  Percent impairment while working due to problem (past 7 days) Week 52 | -10.00 (23.170) | -20.00 (42.426)
  Percent impairment while working due to problem (past 7 days) Week 80: number analyzed (Participants) | 21 | 0
  Percent impairment while working due to problem (past 7 days) Week 80 | -14.76 (26.385) |
  Percent overall work impairment due to problem (past 7 days) Week 4: number analyzed (Participants) | 17 | 15
  Percent overall work impairment due to problem (past 7 days) Week 4 | -9.63 (22.495) | -2.34 (14.807)
  Percent overall work impairment due to problem (past 7 days) Week 8: number analyzed (Participants) | 13 | 13
  Percent overall work impairment due to problem (past 7 days) Week 8 | -11.32 (18.505) | -4.38 (17.568)
  Percent overall work impairment due to problem (past 7 days) Week 16: number analyzed (Participants) | 15 | 14
  Percent overall work impairment due to problem (past 7 days) Week 16 | -10.26 (33.296) | 5.34 (22.063)
  Percent overall work impairment due to problem (past 7 days) Week 28: number analyzed (Participants) | 16 | 4
  Percent overall work impairment due to problem (past 7 days) Week 28 | -15.98 (23.077) | -8.85 (11.722)
  Percent overall work impairment due to problem (past 7 days) Week 52: number analyzed (Participants) | 16 | 2
  Percent overall work impairment due to problem (past 7 days) Week 52 | -12.61 (27.576) | -22.50 (45.962)
  Percent overall work impairment due to problem (past 7 days) Week 80: number analyzed (Participants) | 14 | 0
  Percent overall work impairment due to problem (past 7 days) Week 80 | -14.36 (30.691) |
  Percent activity impairment due to problem (past 7 days) Week 4: number analyzed (Participants) | 61 | 66
  Percent activity impairment due to problem (past 7 days) Week 4 | -11.97 (22.122) | 2.42 (24.310)
  Percent activity impairment due to problem (past 7 days) Week 8: number analyzed (Participants) | 57 | 61
  Percent activity impairment due to problem (past 7 days) Week 8 | -11.58 (24.985) | 1.97 (16.413)
  Percent activity impairment due to problem (past 7 days) Week 16: number analyzed (Participants) | 55 | 62
  Percent activity impairment due to problem (past 7 days) Week 16 | -14.36 (25.222) | 0.65 (18.980)
  Percent activity impairment due to problem (past 7 days) Week 28: number analyzed (Participants) | 54 | 22
  Percent activity impairment due to problem (past 7 days) Week 28 | -11.67 (25.826) | 2.73 (23.941)
  Percent activity impairment due to problem (past 7 days) Week 52: number analyzed (Participants) | 57 | 12
  Percent activity impairment due to problem (past 7 days) Week 52 | -11.23 (25.360) | 0.00 (15.374)
  Percent activity impairment due to problem (past 7 days) Week 80: number analyzed (Participants) | 55 | 0
  Percent activity impairment due to problem (past 7 days) Week 80 | -11.09 (24.166) |

22. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment Questionnaire (WPAI), by Visit in Patients From BAT Group Who Cross Over to Ruxolitinib After Crossover
Description: as for outcome 21
Time Frame: Baseline (last assessment before cross over), Week 4, 8, 16, 24, 28 and 52 after cross-over
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Best Available Therapy (BAT)
Number analyzed (Participants) | 58
Percent
  Percent work time missed due to problem (past 7 days) Week +4: number analyzed (Participants) | 13
  Percent work time missed due to problem (past 7 days) Week +4 | -7.45 (28.102)
  Percent work time missed due to problem (past 7 days) Week +8: number analyzed (Participants) | 13
  Percent work time missed due to problem (past 7 days) Week +8 | -3.90 (33.237)
  Percent work time missed due to problem (past 7 days) Week +16: number analyzed (Participants) | 10
  Percent work time missed due to problem (past 7 days) Week +16 | -2.66 (40.422)
  Percent work time missed due to problem (past 7 days) Week +24: number analyzed (Participants) | 9
  Percent work time missed due to problem (past 7 days) Week +24 | -1.67 (5.000)
  Percent work time missed due to problem (past 7 days) Week +28: number analyzed (Participants) | 10
  Percent work time missed due to problem (past 7 days) Week +28 | 7.06 (21.757)
  Percent work time missed due to problem (past 7 days) Week +52: number analyzed (Participants) | 8
  Percent work time missed due to problem (past 7 days) Week +52 | 1.12 (3.175)
  Percent impairment while working due to problem (past 7 days) Week +4: number analyzed (Participants) | 15
  Percent impairment while working due to problem (past 7 days) Week +4 | -5.33 (9.904)
  Percent impairment while working due to problem (past 7 days) Week +8: number analyzed (Participants) | 14
  Percent impairment while working due to problem (past 7 days) Week +8 | -4.29 (11.579)
  Percent impairment while working due to problem (past 7 days) Week +16: number analyzed (Participants) | 12
  Percent impairment while working due to problem (past 7 days) Week +16 | -10.83 (20.207)
  Percent impairment while working due to problem (past 7 days) Week +24: number analyzed (Participants) | 13
  Percent impairment while working due to problem (past 7 days) Week +24 | -6.92 (13.156)
  Percent impairment while working due to problem (past 7 days) Week +28: number analyzed (Participants) | 12
  Percent impairment while working due to problem (past 7 days) Week +28 | -3.33 (23.868)
  Percent impairment while working due to problem (past 7 days) Week +52: number analyzed (Participants) | 10
  Percent impairment while working due to problem (past 7 days) Week +52 | -6.00 (13.499)
  Percent overall work impairment due to problem (past 7 days) Week +4: number analyzed (Participants) | 13
  Percent overall work impairment due to problem (past 7 days) Week +4 | -10.98 (20.249)
  Percent overall work impairment due to problem (past 7 days) Week +8: number analyzed (Participants) | 13
  Percent overall work impairment due to problem (past 7 days) Week +8 | -6.91 (24.416)
  Percent overall work impairment due to problem (past 7 days) Week +16: number analyzed (Participants) | 10
  Percent overall work impairment due to problem (past 7 days) Week +16 | -4.73 (30.167)
  Percent overall work impairment due to problem (past 7 days) Week +24: number analyzed (Participants) | 9
  Percent overall work impairment due to problem (past 7 days) Week +24 | -6.06 (14.099)
  Percent overall work impairment due to problem (past 7 days) Week +28: number analyzed (Participants) | 10
  Percent overall work impairment due to problem (past 7 days) Week +28 | -1.81 (20.220)
  Percent overall work impairment due to problem (past 7 days) Week +52: number analyzed (Participants) | 8
  Percent overall work impairment due to problem (past 7 days) Week +52 | -4.03 (12.712)
  Percent activity impairment due to problem (past 7 days) Week +4: number analyzed (Participants) | 47
  Percent activity impairment due to problem (past 7 days) Week +4 | -10.43 (19.886)
  Percent activity impairment due to problem (past 7 days) Week +8: number analyzed (Participants) | 51
  Percent activity impairment due to problem (past 7 days) Week +8 | -8.63 (20.978)
  Percent activity impairment due to problem (past 7 days) Week +16: number analyzed (Participants) | 51
  Percent activity impairment due to problem (past 7 days) Week +16 | -8.82 (21.877)
  Percent activity impairment due to problem (past 7 days) Week +24: number analyzed (Participants) | 51
  Percent activity impairment due to problem (past 7 days) Week +24 | -6.47 (25.363)
  Percent activity impairment due to problem (past 7 days) Week +28: number analyzed (Participants) | 49
  Percent activity impairment due to problem (past 7 days) Week +28 | -6.94 (26.395)
  Percent activity impairment due to problem (past 7 days) Week +52: number analyzed (Participants) | 40
  Percent activity impairment due to problem (past 7 days) Week +52 | -7.00 (22.781)

23. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: The Patient Global Impression of Change (PGIC) is comprised of a single question intended to measure a patient's perspective of improvement or deterioration over time relative to treatment. The PGIC uses a seven-point scale where one (1) equals very much improved and seven (7) equals very much worse.
Time Frame: Week 4, 8, 16, 28, 40, 52 and 80
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 74 | 75
Participants
  Week 4: number analyzed (Participants) | 68 | 72
  Week 4: Very much improved | 10 | 0
  Week 4: Much improved | 22 | 8
  Week 4: Minimally improved | 21 | 7
  Week 4: No change | 14 | 50
  Week 4: Minimally worse | 1 | 6
  Week 4: Much worse | 0 | 0
  Week 4: Very much worse | 0 | 1
  Week 8: number analyzed (Participants) | 69 | 70
  Week 8: Very much improved | 11 | 1
  Week 8: Much improved | 27 | 14
  Week 8: Minimally improved | 15 | 9
  Week 8: No change | 15 | 35
  Week 8: Minimally worse | 0 | 10
  Week 8: Much worse | 1 | 0
  Week 8: Very much worse | 0 | 1
  Week 16: number analyzed (Participants) | 66 | 69
  Week 16: Very much improved | 18 | 2
  Week 16: Much improved | 25 | 13
  Week 16: Minimally improved | 13 | 12
  Week 16: No change | 8 | 33
  Week 16: Minimally worse | 2 | 4
  Week 16: Much worse | 0 | 5
  Week 16: Very much worse | 0 | 0
  Week 28: number analyzed (Participants) | 66 | 27
  Week 28: Very much improved | 19 | 0
  Week 28: Much improved | 25 | 4
  Week 28: Minimally improved | 12 | 5
  Week 28: No change | 9 | 15
  Week 28: Minimally worse | 1 | 3
  Week 28: Much worse | 0 | 0
  Week 28: Very much worse | 0 | 0
  Week 40: number analyzed (Participants) | 66 | 19
  Week 40: Very much improved | 23 | 0
  Week 40: Much improved | 30 | 7
  Week 40: Minimally improved | 5 | 2
  Week 40: No change | 6 | 10
  Week 40: Minimally worse | 2 | 0
  Week 40: Much worse | 0 | 0
  Week 40: Very much worse | 0 | 0
  Week 52: number analyzed (Participants) | 70 | 14
  Week 52: Very much improved | 27 | 2
  Week 52: Much improved | 28 | 5
  Week 52: Minimally improved | 8 | 1
  Week 52: No change | 5 | 5
  Week 52: Minimally worse | 2 | 1
  Week 52: Much worse | 0 | 0
  Week 52: Very much worse | 0 | 0
  Week 66: number analyzed (Participants) | 67 | 5
  Week 66: Very much improved | 23 | 1
  Week 66: Much improved | 31 | 1
  Week 66: Minimally improved | 6 | 3
  Week 66: No change | 6 | 0
  Week 66: Minimally worse | 1 | 0
  Week 66: Much worse | 0 | 0
  Week 66: Very much worse | 0 | 0
  Week 80: number analyzed (Participants) | 68 | 0
  Week 80: Very much improved | 22 | 0
  Week 80: Much improved | 24 | 0
  Week 80: Minimally improved | 9 | 0
  Week 80: No change | 10 | 0
  Week 80: Minimally worse | 2 | 0
  Week 80: Much worse | 0 | 0
  Week 80: Very much worse | 1 | 0

24. Secondary Outcome: Summary of Patient Global Impression of Change (PGIC), by Visit in Patients From BAT Group Who Cross Over to Ruxolitinib After Crossover
Description: as for outcome 23
Time Frame: Baseline (last assessment before cross over), Week 4, 8, 16, 24, 28, 40, and 52 after cross-over
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Best Available Therapy (BAT)
Number analyzed (Participants) | 58
Participants
  Week +4: number analyzed (Participants) | 52
  Week +4: Very much improved | 10
  Week +4: Much improved | 13
  Week +4: Minimally improved | 13
  Week +4: No change | 16
  Week +4: Minimally worse | 0
  Week +4: Much worse | 0
  Week +8: number analyzed (Participants) | 53
  Week +8: Very much improved | 11
  Week +8: Much improved | 25
  Week +8: Minimally improved | 9
  Week +8: No change | 7
  Week +8: Minimally worse | 1
  Week +8: Much worse | 0
  Week +16: number analyzed (Participants) | 52
  Week +16: Very much improved | 12
  Week +16: Much improved | 28
  Week +16: Minimally improved | 6
  Week +16: No change | 6
  Week +16: Minimally worse | 0
  Week +16: Much worse | 0
  Week +24: number analyzed (Participants) | 50
  Week +24: Very much improved | 19
  Week +24: Much improved | 17
  Week +24: Minimally improved | 5
  Week +24: No change | 8
  Week +24: Minimally worse | 1
  Week +24: Much worse | 0
  Week +28: number analyzed (Participants) | 50
  Week +28: Very much improved | 18
  Week +28: Much improved | 19
  Week +28: Minimally improved | 6
  Week +28: No change | 6
  Week +28: Minimally worse | 1
  Week +28: Much worse | 0
  Week +40: number analyzed (Participants) | 44
  Week +40: Very much improved | 18
  Week +40: Much improved | 15
  Week +40: Minimally improved | 5
  Week +40: No change | 6
  Week +40: Minimally worse | 0
  Week +40: Much worse | 0
  Week +52: number analyzed (Participants) | 42
  Week +52: Very much improved | 17
  Week +52: Much improved | 16
  Week +52: Minimally improved | 6
  Week +52: No change | 3
  Week +52: Minimally worse | 0
  Week +52: Much worse | 0

25. Secondary Outcome: Number of Participants Developing Thrombosis
Description: Proportion of participants developing any arterial or venous thromboembolic event
Time Frame: From randomization to Week 80 for BAT and Week 260 for Ruxolitinib
Population: Safety Set comprised of all randomized participants who received at least one dose of ruxolitinib or BAT.
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 74 | 75
Participants | 0 | 0

26. Post Hoc Outcome: Total Number of Deaths
Description: On-treatment deaths were reported from the day of first dose of study medication to the End of study (End of Treatment +30 days) visit which was Week 260 or prior (+30 days for Rux + crossover) and Week 80 or prior (+30 days for BAT only). Post-treatment deaths were reported following completion study treatment (Week 80 for patients receiving BAT, or Week 260 for patients receiving ruxolitinib) or from the time of premature discontinuation. Patients were followed for survival every three months up to end of study.
Time Frame: Up to Week 260
Population: Safety Set comprised of all randomized participants who received at least one dose of ruxolitinib or BAT.
Measure: Number; unit: Participants
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 74 | 75
Participants
  Death occurring up to 30 days after end of randomised treatment. | 1 | 1
  Death occurring among patients who died after cross over to ruxolitinib (BAT arm only). | 0 | 3
  Death occurring more than 30 days after end of treatment. | 2 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the day of first dose of study medication to the End of study (End of Treatment +30 days) visit which was Week 260 or prior (+30 days for Rux + crossover) and Week 80 or prior (+30 days for BAT only).
Description: Any signs or symptoms that occured from the day of first dose of study medication to the End of study (End of Treatment +30 days) visit which was Week 260 or prior (+30 days for Rux + crossover) and Week 80 or prior (+30 days for BAT only).
Arm/Group | Ruxolitinib | Best Available Therapy | All Crossover Patients
All-Cause Mortality (participants affected / at risk) | 1/74 | 1/75 | 3/58
Serious Adverse Events (participants affected / at risk) | 34/74 | 9/75 | 23/58
Other Adverse Events (participants affected / at risk) | 73/74 | 56/75 | 56/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib (N=74) | Best Available Therapy (N=75) | All Crossover Patients (N=58)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Hyperleukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 2 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 1
Cardiac disorder (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1
Glaucoma (Eye disorders) | 1 | 0 | 0
Retinal artery occlusion (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 1
General physical health deterioration (General disorders) | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 3 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Meningitis (Infections and infestations) | 0 | 1 | 0
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 2
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Pyonephrosis (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0 | 1
Basosquamous carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Blast cell crisis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bone marrow tumour cell infiltration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Juvenile melanoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 1
Uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Vaginal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Facial neuralgia (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Blue toe syndrome (Vascular disorders) | 1 | 0 | 0
Extremity necrosis (Vascular disorders) | 0 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0
Peripheral artery occlusion (Vascular disorders) | 1 | 0 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 1
Venous haemorrhage (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib (N=74) | Best Available Therapy (N=75) | All Crossover Patients (N=58)
Anaemia (Blood and lymphatic system disorders) | 27 | 1 | 19
Leukocytosis (Blood and lymphatic system disorders) | 5 | 4 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 6 | 3
Thrombocytosis (Blood and lymphatic system disorders) | 8 | 3 | 5
Tinnitus (Ear and labyrinth disorders) | 3 | 2 | 3
Vertigo (Ear and labyrinth disorders) | 4 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2 | 4
Abdominal distension (Gastrointestinal disorders) | 5 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 10 | 1 | 8
Abdominal pain upper (Gastrointestinal disorders) | 5 | 3 | 2
Constipation (Gastrointestinal disorders) | 13 | 4 | 8
Diarrhoea (Gastrointestinal disorders) | 7 | 7 | 4
Dyspepsia (Gastrointestinal disorders) | 5 | 2 | 4
Flatulence (Gastrointestinal disorders) | 1 | 1 | 3
Nausea (Gastrointestinal disorders) | 4 | 5 | 3
Vomiting (Gastrointestinal disorders) | 2 | 1 | 4
Asthenia (General disorders) | 8 | 6 | 6
Fatigue (General disorders) | 13 | 6 | 6
Oedema peripheral (General disorders) | 10 | 2 | 6
Pyrexia (General disorders) | 13 | 1 | 7
Bronchitis (Infections and infestations) | 12 | 2 | 2
Cystitis (Infections and infestations) | 10 | 0 | 2
Herpes zoster (Infections and infestations) | 11 | 0 | 8
Influenza (Infections and infestations) | 10 | 4 | 2
Nasopharyngitis (Infections and infestations) | 8 | 2 | 10
Sinusitis (Infections and infestations) | 1 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 5 | 7 | 5
Urinary tract infection (Infections and infestations) | 6 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 9 | 0 | 2
Blood lactate dehydrogenase increased (Investigations) | 2 | 1 | 4
Gamma-glutamyltransferase increased (Investigations) | 5 | 1 | 1
Haematocrit increased (Investigations) | 0 | 5 | 1
Weight decreased (Investigations) | 1 | 4 | 0
Weight increased (Investigations) | 19 | 1 | 9
Decreased appetite (Metabolism and nutrition disorders) | 5 | 4 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 4
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5 | 0 | 5
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 | 3 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 0 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 2 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 1 | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 2 | 4
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 3
Dizziness (Nervous system disorders) | 8 | 5 | 7
Headache (Nervous system disorders) | 13 | 9 | 8
Memory impairment (Nervous system disorders) | 0 | 0 | 4
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 3
Paraesthesia (Nervous system disorders) | 7 | 0 | 2
Depression (Psychiatric disorders) | 5 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 2 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 7
Erythema (Skin and subcutaneous tissue disorders) | 2 | 4 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 6 | 5 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 17 | 7
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 | 0 | 2
Haematoma (Vascular disorders) | 10 | 1 | 4
Hypertension (Vascular disorders) | 15 | 3 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.